CLINICAL TRIAL: NCT04981925
Title: Predictors of Pain Relief From Mindfulness-based Stress Reduction in Multiple Forms of Chronic Pain Patients
Brief Title: Predictors of Pain Relief From Mindfulness-based Stress Reduction (MBSR) in Multiple Forms of Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Todd Favorite, Director, Psychological Clinic, Clinical Associate Professor of Mary A Rackham Institute, Graduate School and Associate Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00187535
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain Syndrome
Keywords: chronic pain; rheumatoid arthritis; fibromyalgia; neuropathy; neuralgia; pain
MeSH Terms: conditions — Chronic Pain; Arthritis, Rheumatoid; Fibromyalgia; Neuralgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MBSR treatment (Experimental)
  Interventions: Behavioral: MBSR treatment

INTERVENTIONS:
Behavioral: MBSR treatment — Participants will complete pre-treatment surveys followed by 8-weekly 2-hour group sessions and one 4-hour "retreat" (may take place virtually or in-person). Participants will also be asked to practice daily formal mindfulness at home using assigned audio recordings of 30-45 minute guided mindfulness exercises. Participants will complete surveys during treatment as well as after treatment and then at 2 months follow-up.

SUMMARY:
The overall objective of this study is to better understand how Mindfulness-based Stress Reduction (MBSR) is the most helpful in terms of management of chronic pain symptoms.

The studies hypothesis is that an Interventional Response Phenotyping study (light phenotyping) can identify individuals with different underlying mechanisms for their pain who thus respond differentially to evidence-based interventions for chronic pain disorders.

DETAILED DESCRIPTION:
Participants enrolled in this study will receive 8 weeks of MBSR therapy and complete surveys at various time points pre-treatment - post treatment.

ELIGIBILITY:
Inclusion criteria for MBSR Study

* Ages 18+
* Any form of self-reported chronic pain (except cancer related pain)

Exclusion criteria for MBSR study

* Unable to speak and write English
* Visual or hearing difficulties that would preclude participation
* Chronic pain from cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
PROMIS physical function 6b | 8 weeks (after MSBR)
  Physical Function 6b questionnaire will assess self-reported capability with 6 qualitatively scaled questions ranked on a 5-point scale, from "without any difficulty" to "unable to do" or "not at all" to "cannot do." The minimum raw summed score is 6 and the maximum score is 30. Lower scores suggest better outcomes.

SECONDARY OUTCOMES:
Change in PROMIS pain intensity, anxiety, pain interference | Baseline (pre-treatment), 8 weeks
  Change from baseline in pain interference (QoL), measured by PROMIS Pain Interference 6a. Measure of the amount of interference pain causes in life; range 6-30; higher is worse
Change in PROMIS pain intensity, anxiety, pain interference | Baseline (pre-treatment), 8 and 12 weeks
  Change from baseline in pain interference (QoL), measured by PROMIS Pain Interference 6a. Measure of the amount of interference pain causes in life; range 6-30; higher is worse
Change in Pain Catastrophizing Scale (PCS) | Baseline (pre-treatment), 8 and 12 weeks
  The PCS is a 13-item questionnaire that inquires about thoughts and feelings a patient experiences when in pain. Responses are recorded on a 5-point Likert scale ("not at all" to "all the time"). A total score is yielded ranging from 0-52. Higher score is associated with worse outcome.
Pain Catastrophizing Score; measured with Pain Catastrophizing Scale | 8 weeks (after MSBR)
  The PCS is a 13-item questionnaire that inquires about thoughts and feelings a patient experiences when in pain. Responses are recorded on a 5-point Likert scale ("not at all" to "all the time"). A total score is yielded ranging from 0-52. Higher score is associated with worse outcome
Change in Chronic Pain Acceptance Questionnaire (CPAQ)-8 | Baseline, 8 weeks (after MSBR)
  CPAQ-8 is an 8-item questionnaire with a score range 0-48 with higher scores indicating better status. Change score is computed by subtracting baseline CPAQ-8 score from score at time of reassessment. Improvement is indicated by change scores with positive values.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Favorite, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No